CLINICAL TRIAL: NCT06123520
Title: Efficacy of Holmium Laser Urethrotomy Versus in Combination With Intralesional Paclitaxel Injection in the Treatment of Urethral Stricture
Brief Title: Laser Visual Internal Urethrotomy With Versus Without Paclitaxel Injection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Younan Ramsis, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endoscopic VIU 01
Record Dates: First submitted 2023-10-27; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Urethral Stricture, Male
Keywords: Urethral stricture; Visual internal urethrotomy; Paclitaxel submucosal injection
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ho-YAG Laser internal urethrotomy (Active Comparator): consists of those who will undergo Ho-YAG laser internal urethrotomy only.
  Interventions: Procedure: Ho-YAG Laser Visual internal urethrotomy
- Ho-YAG Laser internal urethrotomy + Paclitaxel injection (Experimental): those who will undergo Ho-YAG laser internal urethrotomy with circumferential submucosal paclitaxel injection at the stricture site.
  Interventions: Procedure: Ho-YAG Laser Visual internal urethrotomy combined with intralesional submucosal injection of Paclitaxel

INTERVENTIONS:
Procedure: Ho-YAG Laser Visual internal urethrotomy — the operations will be performed by an expert surgeon and operative time will be considered. The procedure will be performed under spinal or general anaesthesia in lithotomy position. Antibiotic will be given just before and 12 h after procedure and continued for next 5 days.
  Normal saline will be used for irrigation during the procedure. A Holmium laser at an energy of 1,200 to 2.000 mJ with a frequency of 10 to 15 Hz will be used By use of a 22 F cystoscope and Ho:YAG laser, the stricture site will be completely incised while sparing healthy mucosa. a fiber will be positioned about 1 mm away from the tissue and the laser will be fired.
  An 18 F silicone Foley catheter will be left in the urethra at the end of the procedure. urethral catheter removal and voiding trial will be given at postoperative Day 7.
  Other Names: Ho-YAG Laser visual internal urethrotomy (VIU)
  Arms: Ho-YAG Laser internal urethrotomy
Procedure: Ho-YAG Laser Visual internal urethrotomy combined with intralesional submucosal injection of Paclitaxel — The investigators will follow the same interversion protocol in the first group then paclitaxel is going to be injected via Williams cystoscopic injection needle (5 F size and 23 G needle size) through the cystoscope after laser ablation of the stricture in the submucosa with an assumed dose of 3.5µg/mm2 (reaching a urethral diameter of 30 Fr and a total length of 2 cm a total dose of 2.2 mg divided along 3 injection is to be injected). the dose is divided at 12,4 and 8 o'clock respectively along the length of the stricture.
  An 18 F silicone Foley catheter will be left in the urethra at the end of the procedure. urethral catheter removal and voiding trial will be given at postoperative Day 7.
  Other Names: Ho-YAG Laser VIU combined with submucosal Paclitaxel injection
  Arms: Ho-YAG Laser internal urethrotomy + Paclitaxel injection

SUMMARY:
To evaluate the outcome of visual internal urethrotomy in treating urethral strictures in males with a holmium: yttrium-aluminium garnet (YAG) laser versus when combined with intralesional injection of paclitaxel.

DETAILED DESCRIPTION:
Urethral strictures are one of the most common reasons for urological admissions. They are associated with urinary tract infections, bladder stones, fistulas, sepsis and possibly renal insufficiency. Minimally invasive surgical approaches are utilized efficiently and safely in the treatment of urethral strictures. Visualized internal urethrotomy VIU, is one of the preferred methods due to the practical and minimally invasive nature of the procedure. One of the alternative approaches is the correction of the stricture using laser energy. The aim of this prospective study is to evaluate the results of YAG laser internal urethrotomy (HIU) in primary urethral strictures versus using laser with intralesional submucosal paclitaxel injection.

It is a prospective study in which patients will be recruited from the outpatient clinic of Demerdash (ain Shams university) hospital, randomized via closed envelope technique into doing VIU alone versus doing VIU with intralesional injection of paclitaxel

After obtaining well informed written consent, all patients will undergo the following

1. Detailed history taking, including medical history, surgical history, and patient complaint according to international prostate symptom score (IPSS) score. A note will be made about the possible etiology of the stricture.
2. Clinical Examination including abdominal, pelvic and genital examination.
3. Laboratory investigations including complete blood count, urine analysis, urine culture and sensitivity test, renal function tests.
4. Radiological investigations including retrograde urethrogram, micturating cystourethrogram and pelvi-abdominal ultrasound.
5. Uroflowmetry

Any active urinary tract infection (UTI) will be treated before surgery with appropriate antibiotics based upon sensitivity test.

All patients will be followed up intraoperatively recording operative time and the need for blood transfusion, postopertively regarding haemoglobin level, total leucocytic count level and the development of fever or not. All patients will be scheduled to remove the catheter at 14 days postoperative and assessment of international prostate symptom score (IPSS) at first day of catheter removal.

Three months and six months postoperative the patients will be followed up for IPSS, Uroflowmetry results and if the patient is retained (could not urinate) or his results were worse than starting results, then cystourethrogram will be asked from him to investigate the possibility of recurrence.

ELIGIBILITY:
Inclusion criteria:

1. Adult male
2. Presence of obstructive symptoms (moderate to severe according to IPSS scoring system i.e. >7)
3. Single urethral (stricture length <1.5 cm) as evident on radiological studies, i.e., retrograde urethrography (RGU) and micturating cystourethrography (MCU).
4. Average flow rate on uroflowmetry less than 10 ml/s

Exclusion criteria used were:

1. Complete obliteration of lumen of urethra on urethroscopy.
2. Multiple strictures.
3. Untreated urinary tract infection.
4. Recurrent Strictures.
5. Prior internal urethrotomy
6. Prior urethroplasty
7. Compromised upper urinary tract (increased kidney functions)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — urethral stricture in males (urethral stricture in females is rare and has other treatment modalities)
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
International prostate symptom score (IPSS) score | at 3, 6 months
  Clinical effectiveness in improving patient reported lower urinary tract symptoms according to IPSS with a score from 0 to 35 by answering 7 questions, each question with a 0 till 5 points with total score from 0 till 35. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
uroflowmetry | at 3, 6 months
  the quantitative assessment of the flow of urine using uroflowmetry with a score higher than 15 ml/sec indicating no obstruction while from 0-10 indicates obstructed flow and between 10 to 15 obstruction is suspected requiring further investigations.

SECONDARY OUTCOMES:
assessment of operative time. | immediately intraoperative.
  assessment of operative time.
assessment of intraoperative bleeding | immediatly postoperative
  amount of blood loss intraoperative with comparing preoperative and postoperative haemoglobin levels and the need of intraoperative blood transfusion.
assessment of postoperative infection. | Patient will be discharged from hospital being 24 hours fever free postoperative.
  All patients will be followed up intraoperatively recording operative time and the need for blood transfusion, postopertively regarding haemoglobin level, total leucocytic count level and the development of fever or not and the time of discharge from hospital to calculate hospital stay time based upon being 24 hours fever free with no bleeding postoperatively or until the correction of such conditions (resolution of fever and stopping the bleeding with correction of haemoglobin level).
assessment of recurrence rate. | at 3 and 6 months postoperative
  if the patient is retained (could not urinate) or his results in IPSS or Uroflowmetry were worse than starting results, then cystourethrogram will be asked from him to investigate the possibility of recurrence of urethral stricture.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed E. Mousa, Assisstant Professor, Study Director — AinShams University
Locations (1):
- Demerdash hospital, Faculty of medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No